CLINICAL TRIAL: NCT01338935
Title: A Phase I, Single-Site, Tri-Institutional, Open-Label, Three-Part, Dose-Escalation Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of CW002 in Healthy Adult Anesthetized Volunteers
Brief Title: Phase I Clinical Trial to Evaluate the Safety, Pharmacokinetics and Efficacy of CW002
Acronym: CW002
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pharmacokinetic stopping criteria for the study were met.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Cynthia Lien, Attending Anesthesiologist, Weill Medical College of Cornell University
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 1005011060
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: CW 002; Phase I trial; safety; efficacy; pharmacokinetics; estimated dose; Neuromuscular Blocking Agents; Treatment Effectiveness; Drug Antagonism
MeSH Terms: interventions — CW 002

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part I (Experimental): Ascending dose tolerance, PK, and estimation of ED95 for CW 002
  Interventions: Drug: CW 002
- Part II (Experimental): Safety, efficacy and PK of increasing bolus doses and infusions of CW 002, and exploration of Neostigmine reversal
  Interventions: Drug: CW 002
- Part III (Experimental): Intubation with CW 002 and Neostigmine reversal
  Interventions: Drug: CW 002

INTERVENTIONS:
Drug: CW 002 — For Cohort 1, subjects receive a single bolus of 0.02 mg/kg CW 002 (i.v.) and neuromuscular function will be allowed to recover spontaneously for at least 5 half-lives.
  For Cohort 2, an estimated ED50 bolus dose of CW 002 (approximately 0.03 mg/kg) will be given i.v. followed by a second bolus of the same dosage*.
  For Cohort 3, an estimated ED 75 bolus dose of CW 002 (approximately 0.04 mg/kg) will be given i.v. followed by a second bolus of the same dosage *.
  For Cohort IV, an estimated ED 90 bolus dose of CW 002 (approximately 0.06 mg/kg) will be given i.v. followed by a second bolus of the same dosage*.
  *For Cohorts 2-4, a second bolus dose will be administered following a minimum of 5 half-lives of CW002 (based on PK data from Cohort 1).
  Arms: Part I
Drug: CW 002 — Subjects receive an initial ascending bolus dose of CW 002 injection, and a second bolus followed by a continuous infusion initiated at the point of 25% recovery of twitch response. Infusion rate will be adjusted to maintain 97%- 99% suppression of twitch, but to avoid complete neuromuscular block. For the first 3 subjects of each cohort, CW 002 will be allowed to recover spontaneously. For the second 3 subjects, reversal will be performed at the appearance of 1st twitch using 0.05 mg/kg neostigmine and 0.01 mg/kg glycopyrrolate.
  Cohort 5- subject receives 2.0x ED95 dose of CW 002, followed by 1.5x ED95 dose and 30 min infusion of 2-10 mcg/kg/min of CW 002
  Cohort 6 - subject receives 3.0x ED95 dose of CW 002, followed by 1.5x ED95 dose and 60 min infusion of 2-10 mcg/kg/min of CW 002
  Cohort 7 - subject receives 4.0x ED95 dose of CW 002, followed by 1.5x ED95 dose and 90 min infusion of 2-10 mcg/kg/min of CW 002
  Bolus doses of ED95 are determined in Part I of the study.
  Arms: Part II
Drug: CW 002 — In Part III, safety, intubation efficacy, and PK will be evaluated in 2 cohorts (Cohorts 8 and 9) of 6 subjects each, who will undergo endotracheal intubation at 60 or 90 seconds after a bolus dose of CW002 injection at 3 to 4 times the ED95. For the first 3 subjects of each cohort, CW 002 will be allowed to recover spontaneously. For the second 3 subjects, reversal will be performed at the appearance of 1st twitch using 0.05 mg/kg neostigmine and 0.01 mg/kg glycopyrrolate.
  Cohort 8 - subject receives 3.0x ED95 dose of CW 002, and intubation attempt is made 90 seconds post-bolus.
  Cohort 9 - subject receives 4.0x ED95 dose of CW 002, and intubation attempt is made 60 seconds post-bolus.
  Arms: Part III

SUMMARY:
The purpose of this study is to test the safety and efficacy of an investigational neuromuscular blocking agent called CW002 and to document its effects on healthy adult volunteers. A neuromuscular blocking agent is a drug that temporarily prevents muscles from moving. CW002 has not yet been approved by the Food and Drug Administration (FDA).

Usually, neuromuscular blocking agents are used together with other drugs that put people completely "asleep". These drugs allow doctors to place a breathing tube in the airway, stop muscles from moving during surgical operations, and allow ventilation (movement of air).

This research is being done because CW002 is expected to act quickly and to provide a muscle block of intermediate (not too long, not too short) duration. The researchers would like to test increasing doses of CW002 that can be given without causing severe side effects. If shown to be both safe and effective, such a compound would be useful in surgical procedures and could improve future anesthetic care.

DETAILED DESCRIPTION:
Neuromuscular blocking agents are especially important in intubation (insertion of breathing tube into the windpipe) because a quick and effective muscle block is needed to promptly complete the process and secure the airway. In addition, being able to rapidly reverse a blocking agent is desirable so that the patient can breathe on his/her own as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female in good health (ASA I) between the ages of 18 and 49 years inclusive, with no concurrent disease or illness. Females must be non pregnant, non lactating, and practicing an acceptable method of birth control (e.g., barrier, oral contraceptive, vasectomized partner, abstinence) or be surgically sterile or post menopausal. A pregnancy test will be performed at Screening and on Day 1 to confirm non-pregnant status of female subjects.
* Weighs between 55 and 95 kg, inclusive, and has a body mass index (BMI) between 18 and 30 kg/m2 (BMI calculated as weight in kg/[height in m]2 )
* Agrees to abstain from taking any dietary supplements or non-prescription drugs (except for multivitamins or as authorized by the Investigator and Medical Monitor) for 3 days prior to Baseline through Follow-Up
* Agrees to abstain from taking any prescription drugs (except as authorized by the Investigator and Medical Monitor) during the 14 days prior to Baseline through Follow-Up
* Agrees to abstain from consuming alcohol-containing beverages for 3 days prior to Baseline through Follow-up
* Is in good health (ASA Class I) based on medical history and clinically acceptable results on the following assessments: physical examination, vital signs, 12 lead ECG, clinical chemistry, hematology/coagulation, and urinalysis. Seated systolic BP must be > 90 mmHg and ≤ 140 mmHg and seated diastolic BP must be > 50 mmHg and ≤ 90 mmHg at Screening and Baseline
* Has no history of cardiovascular, pulmonary, renal, hepatic, central nervous system, or neuromuscular disease, or history of asthma or diabetes (ASA Class I)
* Is able to communicate effectively with study personnel and is considered reliable, willing, and cooperative in terms of compliance with the protocol requirements
* Voluntarily gives written informed consent to participate in the study
* Has available a responsible adult who has agreed to transport the subject home

Exclusion Criteria:

* Has any current acute or chronic disease
* Has a history of any clinically important medical disorder including any of the following: cardiovascular, pulmonary, hepatic, renal, CNS or neuromuscular disease, asthma or diabetes
* Has a history of anaphylaxis, a documented hypersensitivity reaction, or a clinically important idiosyncratic reaction to any drug
* Has a history of neuromuscular junction disease (e.g., myotonic dystrophy, polio, myasthenia gravis, botulism poisoning)
* Has a history of malignant hyperthermia
* Has had recent (within 2 weeks) use of aminoglycoside antibiotics or corticosteroids
* Has a history of sleep apnea
* Has a history of prior anesthetic complications
* Has any history of asthma requiring management for reactive airway disease
* Has a history of an anatomic airway abnormality or indication of an airway abnormality assessed during the Screening airway examination that could interfere with laryngoscopy or tracheal intubation
* Has a history of Human Immunodeficiency Virus (HIV) infection or Acquired Immune Deficiency Syndrome (AIDS), or has a history of viral hepatitis (other than Hepatitis A)
* Has a history of malignancy within the past 5 years, with the exception of successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin and/or localized carcinoma in situ of the cervix
* Has a predisposing condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs or any condition that may confound the PK analyses, particularly hepatic or renal disease
* Has received another investigational drug within 30 days prior to the Screening Visit
* Has a history of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit) and/or evidence of any use within 3 days prior to Baseline
* Has a history or current evidence of abuse of licit or illicit drug substances or a positive urine drug screen for drugs of abuse
* Currently uses tobacco-containing products or has a history of tobacco use within 6 months prior to the Screening Visit
* Has donated blood or plasma within 60 days prior to the Screening Visit
* Has an abnormal bleeding tendency

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the use of CW002 in healthy human volunteers by monitoring changes in ECG, heart rate (HR), mean arterial pressure, plasma histamine levels, clinical laboratory values, and noting the occurrence of adverse events. | 4 weeks

SECONDARY OUTCOMES:
To estimate the ED95 (dose required to produce 95% suppression of neuromuscular activity | 24 hours
  Neuromuscular activity is measured by the mechanomyographic response of the adductor pollicis (a muscle in the hand that functions to move the thumb muscle) to indirect stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Lien, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Belmont MR, Lien CA, Tjan J, Bradley E, Stein B, Patel SS, Savarese JJ. Clinical pharmacology of GW280430A in humans. Anesthesiology. 2004 Apr;100(4):768-73. doi: 10.1097/00000542-200404000-00004. PMID 15087609
- [Background] Donati F. Neuromuscular blocking drugs for the new millennium: current practice, future trends--comparative pharmacology of neuromuscular blocking drugs. Anesth Analg. 2000 May;90(5 Suppl):S2-S6. doi: 10.1097/00000539-200005001-00002. No abstract available. PMID 10809511
- [Background] Kopman AF, Klewicka MM, Neuman GG. An alternate method for estimating the dose-response relationships of neuromuscular blocking drugs. Anesth Analg. 2000 May;90(5):1191-7. doi: 10.1097/00000539-200005000-00036. PMID 10781478
- [Background] Kopman AF, Klewicka MM, Neuman GG. Reexamined: the recommended endotracheal intubating dose for nondepolarizing neuromuscular blockers of rapid onset. Anesth Analg. 2001 Oct;93(4):954-9. doi: 10.1097/00000539-200110000-00030. PMID 11574363
- [Background] Savarese JJ, McGilvra JD, Sunaga H, Belmont MR, Van Ornum SG, Savard PM, Heerdt PM. Rapid chemical antagonism of neuromuscular blockade by L-cysteine adduction to and inactivation of the olefinic (double-bonded) isoquinolinium diester compounds gantacurium (AV430A), CW 002, and CW 011. Anesthesiology. 2010 Jul;113(1):58-73. doi: 10.1097/ALN.0b013e3181dc1b5b. PMID 20526187
- [Background] Viby-Mogensen J, Engbaek J, Eriksson LI, Gramstad L, Jensen E, Jensen FS, Koscielniak-Nielsen Z, Skovgaard LT, Ostergaard D. Good clinical research practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents. Acta Anaesthesiol Scand. 1996 Jan;40(1):59-74. doi: 10.1111/j.1399-6576.1996.tb04389.x. PMID 8904261